CLINICAL TRIAL: NCT03965130
Title: The Effect of Glucagon on Rates of Hepatic Mitochondrial Oxidation and Pyruvate Carboxylase Flux in Man Assessed by Positional Isotopomer NMR Tracer Analysis (PINTA)
Brief Title: The Effect of Glucagon on Rates of Hepatic Mitochondrial Oxidation in Man Assessed by PINTA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0209020997_a; MISP58340 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants
Keywords: Hepatic Glucose Metabolism; Hepatic Mitochondrial Oxidation; PINTA; Glucagon
MeSH Terms: conditions — Pinta | interventions — Glucagon

STUDY DESIGN:
Intervention Model Description: Each participant will participate in two studies: one without and one with a 3 hour infusion of glucagon during the PINTA study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucagon (Experimental): Participants will receive glucagon during the PINTA study
  Interventions: Biological: Glucagon
- Control (Experimental): The same participants will not receive glucagon during the PINTA study
  Interventions: Other: Control Study

INTERVENTIONS:
Biological: Glucagon — PINTA study with glucagon
  Other Names: hormone study
  Arms: Glucagon
Other: Control Study — The same participants will not receive glucagon during the PINTA study
  Other Names: No glucagon
  Arms: Control

SUMMARY:
It is well established that alterations in the portal vein insulin:glucagon ratio play a major role in the dysregulated hepatic glucose metabolism in type 2 diabetes but the molecular mechanism by which glucagon promotes alterations in hepatic glucose production and mitochondrial oxidation remain poorly understood. This is borne out of the fact that both glucagon agonists and antagonists are being developed to treat type 2 diabetes with unclear mechanisms of action.

This study will directly assess rates of mitochondrial oxidation and pyruvate carboxylase flux for the first time in humans using PINTA analysis as well as the effects of glucagon. The results will have important implications for the possibility of intervening in the pathogenesis of non alcoholic fatty liver and type 2 diabetes via chronic dual GLP-1/glucagon receptor antagonism and provide an important rationale for why a dual agonist may be more efficacious for treatment of non alcoholic fatty liver and T2D than GLP-1 alone.

DETAILED DESCRIPTION:
Objectives:

To examine rates of hepatic mitochondrial oxidation in healthy volunteers with liver lipid less than 2%.

To examine the effects of glucagon on hepatic glucose and fat metabolism in vivo, this study will apply a novel Positional Isotopomer NMR Tracer Analysis (PINTA) method to quantify rates of hepatic mitochondrial oxidation and pyruvate carboxylase flux, which has been cross-validated in awake rodents and humans (Perry et al. Nature Communications 2017). Preliminary rodent studies have found that glucagon stimulates intrahepatic lipolysis through an InsP3R-I-dependent process, leading to increases in hepatic acetyl-CoA content, which allosterically activates pyruvate carboxylase activity and flux, and that this phenomenon explains its acute, transcription-independent effect to acutely stimulate hepatic gluconeogenesis in vivo (unpublished results). In addition, using PINTA analysis it has been shown that glucagon stimulates hepatic mitochondrial oxidation through calcium signaling in awake mice, and that this process can be exploited by short-term continuous glucagon treatment leading to two-fold increases in hepatic mitochondrial fat oxidation, which in turn results in large reductions in hepatic steatosis and marked improvements in glucose tolerance through reversal of hepatic insulin resistance in a high fat fed rat model of non alcoholic fatty liver.

Hypothesis:

1. A physiological increase in plasma glucagon concentrations will promote a significant increase in rates of hepatic mitochondrial oxidation in healthy humans.

3. A physiological increase in plasma glucagon concentrations will promote a significant increase in rates of hepatic pyruvate carboxylase flux in healthy humans.

4. A physiological increase in plasma glucagon concentrations will promote a significant increase in rates of 13C4 β-hydroxybutyrate turnover (hepatic ketogenesis) in healthy humans.

Study Design - Clinical Plan:

The effects of a physiological increase in plasma glucagon on rates of hepatic mitochondrial oxidation and pyruvate carboxylase flux will be examined in a group of up to 12 healthy participants (ages 21-65) using Positional Isotopomer NMR Tracer Analysis (PINTA) (Perry et al. Nature Communication 2017). Briefly rates of hepatic mitochondrial oxidation and hepatic pyruvate carboxylase flux will be assessed in 12 healthy overnight fasted participants by PINTA after a three-hour infusion of glucagon or saline. The glucagon infusion will be designed to increase peripheral and portal vein plasma glucagon concentrations 3-4 fold. The effects of a physiological increase in plasma glucagon on rates of hepatic ketogenesis will also be assessed using an infusion of 13C4 β-betahydroxybutyrate (Perry et al. Cell Metabolism 2017).

Rates of hepatic pyruvate carboxylase flux /citrate synthase flux by PINTA: Participants (n=12) will be studied by PINTA under 2 conditions: 1) following an overnight fast and a 3 hour saline infusion (Control), 2) following an overnight fast and a 3 hour glucagon infusion. Briefly, after collection of baseline blood samples a 3 hour infusion of tracers as described below will be started. Relative rates of pyruvate carboxylase to citrate synthesis flux will be assessed using a constant infusion of [3-13C] lactate and rates of glucose production will be measured using an infusion of [2H7]glucose (Perry et al. Nature Communication 2017). Rates of hepatic ketogenesis will be measured using a constant infusion of [3C β-hydroxybutyrate as previously described (Perry et al. Cell Metabolism 2017).

Whole body energy expenditure and the respiratory quotient will be assessed by indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non smoking
* Taking no medications except birth control

Exclusion Criteria:

* Any systemic or organ disease
* Smoking
* Taking any drug or medications other than birth control (women)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kitt F Petersen, MD, Principal Investigator — Professor
Locations (1):
- Yale Hospital reserach Unit / YCCI, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Final data to be shared with study sponsor

RESULTS

PARTICIPANT FLOW:
Groups:
- Glucagon: Participants will receive glucagon or saline during the PINTA study
  Glucagon: PINTA study with or without glucagon
Period: Overall Study
Arm/Group | Glucagon
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Glucagon
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Hepatic mitochondrial function [Mean (Standard Deviation); unit: micromol per min] | 149 (49)

OUTCOME MEASURES:

1. Primary Outcome: Rates of Hepatic Mitochondrial Oxidation
Description: Rates of pyruvate carboxylase flux and citrate synthesis flux will be assessed using GC/MS and NMR analyses of plasma glucose 13C enrichments after the [3-13C]lactate infusion
Time Frame: 5 hours
Population: Each arm is comprised of the same 10 participants from the crossover design.
Measure: Mean (Standard Error); unit: micromol/min
Groups:
- Saline: Participants will receive glucagon or saline during the PINTA study
  Glucagon: PINTA study with or without glucagon
Arm/Group | Glucagon | Saline
Number analyzed (Participants) | 10 | 10
micromol/min | 262 (33) | 149 (15)

ADVERSE EVENTS:
Time Frame: Each participant completed the two studies over a period of 4 weeks. Each was a one-time study with PINTA tracer infusions with or with our a glucagon infusion added. Adverse events were monitored throughout both the first study and the second study.
Description: Adverse events would be IV site irritation, nausea due to the glucagon administration.
Groups:
- Glucagon: Participants will receive glucagon in the PINTA study
Arm/Group | Glucagon | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03965130/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT03965130/ICF_002.pdf